CLINICAL TRIAL: NCT02279849
Title: Multi-level Communications and Access Strategies to Improve the Food Environment:B'More Healthy: Retailer Rewards (BHRR)
Brief Title: Multi-level Communications and Access Strategies to Improve the Food Environment
Acronym: BHRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Joel Gittelsohn, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: NIH110547
Record Dates: First submitted 2014-02-18; First posted 2014-10-31 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Obesity
Keywords: multi-level intervention; price discounts; communication; low income population; dietary intervention; obesity prevention; store-based intervention
MeSH Terms: conditions — Obesity; Communication | interventions — Costs and Cost Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Communications (Experimental): These 6 stores received the communications intervention. Communications materials were developed for each program phase; 1) Healthier Drinks, 2) Healthier Essentials, and 3) Healthier Snacks. Each phase's materials included posters, recipe cards, educational handouts, shelf talkers, price tags, door signs, educational displays, and promotional giveaways (i.e., drink tumblers, re-usable shopping bags) to encourage healthy food purchasing and consumption. Stores receiving the communications intervention also received either a small refrigerator or freezer to help provide the environmental supports needed to stock perishable fruits and vegetables.
  Interventions: Other: Communications
- Control (No Intervention): These 6 stores received no intervention.
- Pricing (Experimental): These 6 stores received a pricing intervention. 10-30% with discounts for specific foods contingent on price elasticity of demand, initial wholesale price, and projected store-level sales. Items were given the minimum discount needed to increase store supply and consumer demand. For example, brand name frozen vegetables were discounted 30% at the wholesaler, in order to provide the storeowner with enough incentive to stock the item. The % discount passed from the storeowner to the consumer was ultimately a decision made by the storeowner, but was suggested to be at least 50% in order to increase consumer demand. Discounts were automatically applied at wholesaler registers to stores receiving the pricing intervention.
  Interventions: Other: Pricing
- Combined (Communications & Pricing) (Experimental): These 6 stores received communications materials as well as pricing incentives as intervention (see Communications & Pricing Arms Descriptions).
  Interventions: Other: Combined (Communications & Pricing)

INTERVENTIONS:
Other: Communications — Communication materials were used to promote healthier items to consumers in corner stores.
  Arms: Communications
Other: Pricing — The pricing incentives were used to help promote sales of healthier food items.
  Arms: Pricing
Other: Combined (Communications & Pricing) — Communications with Pricing incentives were used to promote the sale/consumption of healthier foods.
  Arms: Combined (Communications & Pricing)

SUMMARY:
The overarching goal of B'More Healthy Retail Rewards (BHRR) is to develop, implement, and evaluate a pilot multi-level communications and pricing intervention to improve access to and consumption of healthy foods in low-income areas of Baltimore City, Maryland. BHRR has three primary aims: (1) to conduct formative research with representatives of multiple levels of the Baltimore food environment (i.e., local wholesalers, retail food store owners, and consumers) in order to select key foods for promotion, and determine appropriate communications and healthy food price reduction strategies, (2) to pilot the multi-level program with 2 local wholesale stores, and 24 small corner stores and their customers, and assess program implementation through detailed process evaluation, and (3) to assess impact of multilevel health communications and pricing strategies, combined and separately, on consumer dietary patterns and food source use, food purchasing behaviors, psychosocial variables, food security, and individual weight and height.

DETAILED DESCRIPTION:
Innovative and culturally appropriate multilevel health communications interventions are desperately needed to address the chronic disease epidemic in high-risk populations, such as low-income urban African Americans. However, the vast majority of communications strategies have focused on educating individual consumers about healthy food choices, while in poor urban settings the lower availability of affordable healthy food choices greatly limits the impact of these messages. The study team worked with 1 wholesaler and 24 small retail food stores to develop and test novel strategies in Baltimore, Maryland, including: 1) multilevel health communications alone directed at wholesalers, retailers and low-income African American consumers intended to enhance willingness to stock and/or purchase healthy foods; 2) pricing strategies (performance based allowances) directed at wholesalers and retailers to increase their stocking of healthy foods at reduced prices; and 3) combined health communications and pricing strategies. Intervention strategies were tailored to meet the needs of the target populations based on formative research and stakeholder input. This research study is based on significant field experience in this setting, including the development of evaluation tools to assess change in stocking and pricing of key foods (at the store level), and psychosocial factors, dietary intake, and food purchasing behaviors (at the consumer level). There are 3 main study aims:

1. Formative research with representatives of multiple levels of the Baltimore food environment (i.e., local wholesalers and retail food store owners) in order to select key foods for promotion, determine appropriate communication strategies (e.g., messages, channels, materials) for each level, and select the most appropriate pricing approach (i.e., performance based allowance structure and stipulations).
2. Pilot the multilevel program with three wholesalers and 24 food stores (6 control, 6 health communications only, 6 pricing only, 6 combined), and assess program implementation through detailed process evaluation.
3. Assess impact of the pilot program on a) the stocking, pricing, marketing, and sales volume of promoted foods at wholesale and retail levels, and b) food purchasing behaviors and associated psychosocial variables (i.e., self-efficacy, intentions, perceived cost) at the consumer level (final sample n=12 consumers/store, 288 total).

The proposed research seeks to develop effective, multilevel communication strategies to improve diet and reduce risk for diet-related chronic diseases. The study team anticipates this design will demonstrate the value of a multi-pronged and multilevel health communications approach to obesity and chronic disease prevention, and will lead to a large-scale trial and informed policies designed to improve food availability and affordability in low-income urban settings.

ELIGIBILITY:
Inclusion Criteria:

* 21 yrs of age and a regular customer at participating corner store.

Exclusion Criteria:

* Under 21 years of age and not a regular customer of participating store.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Healthy food purchasing and related-psychosocial factors | Up to 8 months
  We analyzed the average change in consumer purchase of promoted foods and related consumer psychosocial variables across treatment groups from baseline and post-intervention by examine intervention effects by analyzing the change variable obtained by subtracting the pretest score from post-test score (exploratory analysis); and 2) conduct confirmatory testing of intervention effects using ANOVA and mixed models.

SECONDARY OUTCOMES:
Consumer dietary intake and consumption of promoted foods | Up to 8 months
  We analyzed the average change in consumer dietary intake and consumption of promoted foods across treatment groups from baseline and post-intervention by examine intervention effects by analyzing the change variable obtained by subtracting the pretest score from post-test score (exploratory analysis); and 2) conduct confirmatory testing of intervention effects using ANOVA and mixed models.

OTHER OUTCOMES:
Store owner psychosocial variables to stock/sell promoted foods | Up to 8 months
  We analyzed the average change in store owner psychosocial variables to stock/sell promoted foods across treatment groups from baseline and post-intervention examine intervention effects by analyzing the change variable obtained by subtracting the pretest score from post-test score (exploratory analysis); and 2) conduct confirmatory testing of intervention effects using ANOVA and mixed models.
Sales of promoted foods | Up to 8 months
  We analyzed the average change in store sales of promoted foods across treatment groups from baseline and post-intervention examine intervention effects by analyzing the change variable obtained by subtracting the pretest score from post-test score (exploratory analysis); and 2) conduct confirmatory testing of intervention effects using ANOVA and mixed models.
Consumer Body Mass Index (BMI) | Up to 11 months
  Average change in consumer consumer BMI across treatment groups from baseline and post-intervention.
Household food security, food assistance, health beliefs, socio-demographics | Up to 11 months
  We analyzed the average change in consumer household food security, food assistance, health beliefs, socio-demographics across treatment groups from baseline and post-intervention examine intervention effects by analyzing the change variable obtained by subtracting the pretest score from post-test score (exploratory analysis); and 2) conduct confirmatory testing of intervention effects using ANOVA and mixed models.
Wholesaler sales of promoted foods | Up to 8 months
  We analyzed the average change in wholesaler sales of promoted foods across treatment groups from baseline and post-intervention examine intervention effects by analyzing the change variable obtained by subtracting the pretest score from post-test score (exploratory analysis); and 2) conduct confirmatory testing of intervention effects using ANOVA and mixed models.
Process Evaluation | Up to 8 months
  Assessing the reach, dose, and fidelity of all intervention components from our post data collection instruments.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Budd N, Cuccia A, Jeffries JK, Prasad D, Frick KD, Powell L, Katz FA, Gittelsohn J. B'More Healthy: Retail Rewards--design of a multi-level communications and pricing intervention to improve the food environment in Baltimore City. BMC Public Health. 2015 Mar 24;15:283. doi: 10.1186/s12889-015-1616-6. PMID 25885923
- See also: website detailing ongoing projects to improve the food environment — http://healthystores.org/